CLINICAL TRIAL: NCT03577197
Title: Southeast Netherlands Advanced Breast Cancer Registry
Brief Title: Southeast Netherlands Advanced Metastatic Breast Cancer Registry
Acronym: SONABRE
Status: Recruiting | Type: Observational
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: Novartis (Industry); Pfizer (Industry); Roche Pharma AG (Industry); Eli Lilly and Company (Industry); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Eisai Inc. (Industry); Daiichi Sankyo (Industry); AstraZeneca (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, V.C.G. Tjan-Heijnen, Professor of medical oncology, Academisch Ziekenhuis Maastricht
Other Study IDs: MUMC-MO-2015-01
Record Dates: First submitted 2018-06-11; First posted 2018-07-05 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: Breast neoplasms; Neoplasm Metastasis; Registry
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Southeast Netherlands Advanced Breast Cancer (SONABRE) Registry is a real life multi-center study. The registry aims to include all patients diagnosed with advanced breast cancer as of 2007 in 11 hospitals in the Netherlands. Data on patient, tumor and treatment characteristics are collected retrospectively from electronic medical files by trained registry clerks.

DETAILED DESCRIPTION:
This SONABRE registry is an ongoing observational cohort study aiming at the inclusion of all patients aged ≥18 years and diagnosed with advanced breast cancer since 2007 in 11 hospitals in the Southeast of the Netherlands. Patients with de novo or recurrent advanced breast cancer were identified from the hospital-based management information systems. Specially trained registration clerks retrospectively collected data from the medical files of the patients based on extensive medical chart review. Information was collected about patient and tumour characteristics, type of treatment (surgery, radiotherapy and systemic treatment, both neo-adjuvant, adjuvant and palliative), palliative treatment changes due to adverse events, hospitalization, comorbidities and outcomes (progression and death). The SONABRE Registry has already been effectively used to perform real-life studies on the use, safety and (cost-)effectiveness of various systemic treatments used in patients diagnosed with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with de novo or recurrent advanced breast cancer since 2007
* Diagnosed with or treated for advanced breast cancer in one of the participating hospitals
* Participating hospitals (period of inclusion): Maastricht UMC+ (2007-2025), Zuyderland hospitals Sittard/Heerlen (2007-2025), Amphia Hospital Breda (2013-2025), Catharina Hospital Eindhoven (2007-2025), Elkerliek Hospital Helmond (2010-2025), Maxima Medical Center Veldhoven/Eindhoven (2007-2025), Jeroen Bosch Hospital Den Bosch (2013-2025), Laurentius Hospital Roermond (2007-2025), St. Annaziekenhuis Geldrop (2007-2025), St. Elisabeth Hospital Tilburg (2007-2009), St. Jans Gasthuis Weert (2007-2025), VieCuri Medical Center Venlo/Venray (2013-2025), all in the Netherlands.
* Hospitals (and periods) were eligible for inclusion if (distant) registration from Maastricht UMC+ was possible.
* The inclusion period may be prolonged after 2025.

Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patient diagnosed with advanced breast cancer since 2007 in 11 hospitals in the Netherlands. No patients are being excluded. Also patients with no systemic / active anti-tumour therapy for advanced breast cancer will be included. The SONABRE Registry includes 11 hospitals: 1 academic, 7 teaching and 3 general hospitals. The Netherlands counts 114 hospitals, including 8 academic, 25 teaching, 58 general and 23 categorical hospitals.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment pattern | up to 13 years
  Treatment pattern per palliative treatment line; proportion of patients receiving chemotherapy, chemotherapy plus targeted therapy, endocrine therapy, endocrine therapy plus targeted therapy or targeted therapy alone

SECONDARY OUTCOMES:
OS | up to 13 years
  Overall survival
PFS | up to 13 years
  Progression-free survival per systemic agent or palliative treatment line
ICER | up to 13 years
  Incremental cost-effectiveness ratio per QALY (quality-adjusted life year) gained of a new systemic drug compared with standard care
QoL | upt to 13 years
  Quality of life; health state utility score calculated from the EQ-5D questionnaire
Costs | up to 13 years
  Costs of advanced breast cancer care from a hospital perspective

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple hospitals in the Netherlands (see Eligibility), Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lobbezoo DJ, van Kampen RJ, Voogd AC, Dercksen MW, van den Berkmortel F, Smilde TJ, van de Wouw AJ, Peters FP, van Riel JM, Peters NA, de Boer M, Peer PG, Tjan-Heijnen VC. Prognosis of metastatic breast cancer: are there differences between patients with de novo and recurrent metastatic breast cancer? Br J Cancer. 2015 Apr 28;112(9):1445-51. doi: 10.1038/bjc.2015.127. Epub 2015 Apr 16. PMID 25880008
- [Result] Lobbezoo DJ, van Kampen RJ, Voogd AC, Dercksen MW, van den Berkmortel F, Smilde TJ, van de Wouw AJ, Peters FP, van Riel JM, Peters NA, de Boer M, Borm GF, Tjan-Heijnen VC. Prognosis of metastatic breast cancer subtypes: the hormone receptor/HER2-positive subtype is associated with the most favorable outcome. Breast Cancer Res Treat. 2013 Oct;141(3):507-14. doi: 10.1007/s10549-013-2711-y. Epub 2013 Oct 9. PMID 24104881
- [Result] Lobbezoo D, Truin W, Voogd A, Roumen R, Vreugdenhil G, Dercksen MW, van den Berkmortel F, Smilde T, van de Wouw A, van Kampen R, van Riel J, Peters N, Peer P, Tjan-Heijnen VC. The role of histological subtype in hormone receptor positive metastatic breast cancer: similar survival but different therapeutic approaches. Oncotarget. 2016 May 17;7(20):29412-9. doi: 10.18632/oncotarget.8838. PMID 27121067
- [Result] Lobbezoo DJ, van Kampen RJ, Voogd AC, Dercksen MW, van den Berkmortel F, Smilde TJ, van de Wouw AJ, Peters FP, van Riel JM, Peters NA, de Boer M, Peer PG, Tjan-Heijnen VC. In real life, one-quarter of patients with hormone receptor-positive metastatic breast cancer receive chemotherapy as initial palliative therapy: a study of the Southeast Netherlands Breast Cancer Consortium. Ann Oncol. 2016 Feb;27(2):256-62. doi: 10.1093/annonc/mdv544. Epub 2015 Nov 16. PMID 26578730
- [Result] van Kampen RJW, Ramaekers BLT, Lobbezoo DJA, de Boer M, Dercksen MW, van den Berkmortel F, Smilde TJ, van de Wouw AJ, Peters FPJ, van Riel JMG, Peters NAJB, Tjan-Heijnen VCG, Joore MA. Real-world and trial-based cost-effectiveness analysis of bevacizumab in HER2-negative metastatic breast cancer patients: a study of the Southeast Netherlands Breast Cancer Consortium. Eur J Cancer. 2017 Jul;79:238-246. doi: 10.1016/j.ejca.2017.01.027. Epub 2017 Feb 27. PMID 28245951
- [Result] Knapen LM, Geurts SME, Ibragimova KIE, Croes S, Vriens BEPJ, van den Berkmortel FWPJ, Dercksen MW, van de Wouw AJ, Pepels MJAE, de Fallois AOJ, Lobbezoo DJA, de Boer M, Tjan-Heijnen VCG. A real-life study on the implementation and effectiveness of exemestane plus everolimus per hospital type in patients with advanced breast cancer. A study of the Southeast Netherlands Advanced Breast Cancer registry. Breast. 2019 Apr;44:46-51. doi: 10.1016/j.breast.2019.01.001. Epub 2019 Jan 4. PMID 30641299
- [Result] Pouwels XGLV, Geurts SME, Ramaekers BLT, Erdkamp F, Vriens BEPJ, Aaldering KNA, van de Wouw AJ, Dercksen MW, Smilde TJ, Peters NAJB, Riel JMV, Pepels MJ, Heijnen-Mommers J, Joore MA, Tjan-Heijnen VCG, de Boer M. The relative effectiveness of eribulin for advanced breast cancer treatment: a study of the southeast Netherlands advanced breast cancer registry. Acta Oncol. 2020 Jan;59(1):82-89. doi: 10.1080/0284186X.2019.1670356. Epub 2019 Oct 4. PMID 31583931
- [Result] Schneider PP, Pouwels XGLV, Passos VL, Ramaekers BLT, Geurts SME, Ibragimova KIE, de Boer M, Erdkamp F, Vriens BEPJ, van de Wouw AJ, den Boer MO, Pepels MJ, Tjan-Heijnen VCG, Joore MA. Variability of cost trajectories over the last year of life in patients with advanced breast cancer in the Netherlands. PLoS One. 2020 Apr 9;15(4):e0230909. doi: 10.1371/journal.pone.0230909. eCollection 2020. PMID 32271794
- [Result] Pouwels XGLV, Ramaekers BLT, Geurts SME, Erdkamp F, Vriens BEPJ, Aaldering KNA, van de Wouw AJ, Dercksen MW, Smilde TJ, Peters NAJB, van Riel JMGH, Pepels MJ, Heijnen-Mommers J, Tjan-Heijnen VCG, de Boer M, Joore MA. An economic evaluation of eribulin for advanced breast cancer treatment based on the Southeast Netherlands advanced breast cancer registry. Acta Oncol. 2020 Sep;59(9):1123-1130. doi: 10.1080/0284186X.2020.1775289. Epub 2020 Jun 16. PMID 32544366
- [Result] Claessens AKM, Ramaekers BLT, Lobbezoo DJA, van Kampen RJW, de Boer M, van de Wouw AJ, Dercksen MW, Geurts SME, Joore MA, Tjan-Heijnen VCG. Quality of life in a real-world cohort of advanced breast cancer patients: a study of the SONABRE Registry. Qual Life Res. 2020 Dec;29(12):3363-3374. doi: 10.1007/s11136-020-02604-4. Epub 2020 Aug 20. PMID 32816222
- [Result] Ibragimova KIE, Geurts SME, Croes S, Erdkamp F, Heijns JB, Tol J, Vriens BEPJ, Aaldering KNA, Dercksen MW, Pepels MJAE, Peters NAJB, van de Winkel L, Tilli DJP, Vriens IJH, de Boer M, Tjan-Heijnen VCG. Survival before and after the introduction of pertuzumab and T-DM1 in HER2-positive advanced breast cancer, a study of the SONABRE Registry. Breast Cancer Res Treat. 2021 Jul;188(2):571-581. doi: 10.1007/s10549-021-06178-8. Epub 2021 Mar 20. PMID 33743103
- [Result] Meegdes M, Ibragimova KIE, Lobbezoo DJA, Vriens IJH, Kooreman LFS, Erdkamp FLG, Dercksen MW, Vriens BEPJ, Aaldering KNA, Pepels MJAE, van de Winkel LMH, Tol J, Heijns JB, van de Wouw AJ, Peters NAJB, Hochstenbach-Waelen A, Smidt ML, Geurts SME, Tjan-Heijnen VCG. The initial hormone receptor/HER2 subtype is the main determinator of subtype discordance in advanced breast cancer: a study of the SONABRE registry. Breast Cancer Res Treat. 2022 Apr;192(2):331-342. doi: 10.1007/s10549-021-06472-5. Epub 2022 Jan 13. PMID 35025003
- [Result] Meegdes M, Geurts SME, Erdkamp FLG, Dercksen MW, Vriens BEPJ, Aaldering KNA, Pepels MJAE, van de Winkel LMH, Teeuwen NJA, de Boer M, Tjan-Heijnen VCG. The implementation of CDK 4/6 inhibitors and its impact on treatment choices in HR+/HER2- advanced breast cancer patients: A study of the Dutch SONABRE Registry. Int J Cancer. 2022 Jan 1;150(1):124-131. doi: 10.1002/ijc.33785. Epub 2021 Sep 14. PMID 34460112
- [Result] Schmitz RSJM, Geurts SME, Ibragimova KIE, Tilli DJP, Tjan-Heijnen VCG, de Boer M. Healthcare Use during the Last Six Months of Life in Patients with Advanced Breast Cancer. Cancers (Basel). 2021 Oct 20;13(21):5271. doi: 10.3390/cancers13215271. PMID 34771434
- [Result] Ibragimova KIE, Geurts SME, Meegdes M, Erdkamp F, Heijns JB, Tol J, Vriens BEPJ, Dercksen MW, Aaldering KNA, Pepels MJAE, van de Winkel L, Peters NAJB, Teeuwen-Dedroog NJA, Vriens IJH, Tjan-Heijnen VCG. Outcomes for the first four lines of therapy in patients with HER2-positive advanced breast cancer: results from the SONABRE registry. Breast Cancer Res Treat. 2023 Apr;198(2):239-251. doi: 10.1007/s10549-022-06832-9. Epub 2023 Jan 12. PMID 36635428
- [Result] Ibragimova KIE, Geurts SME, Laczko D, Meegdes M, Erdkamp F, Heijns JB, Tol J, Vriens BEPJ, Aaldering KNA, Dercksen MW, Pepels MJAE, Peters NAJB, van de Winkel LMH, van de Wouw AJ, de Fallois A, van Kats MACE, Tjan-Heijnen VCG. Trastuzumab Resistance in Patients With HER2-Positive Advanced Breast Cancer: Results From the SONABRE Registry. Clin Breast Cancer. 2024 Feb;24(2):103-111. doi: 10.1016/j.clbc.2023.10.009. Epub 2023 Nov 2. PMID 38007349
- [Result] Meegdes M, Geurts SME, Erdkamp FLG, Dercksen MW, Vriens BEPJ, Aaldering KNA, Pepels MJAE, van de Winkel LMH, Peters NAJB, Tol J, Heijns JB, van de Wouw AJ, de Fallois AJO, van Kats MACE, Tjan-Heijnen VCG. Real-world time trends in overall survival, treatments and patient characteristics in HR+/HER2- metastatic breast cancer: an observational study of the SONABRE Registry. Lancet Reg Health Eur. 2023 Jan 6;26:100573. doi: 10.1016/j.lanepe.2022.100573. eCollection 2023 Mar. PMID 36895447
- [Result] Geurts SME, Ibragimova KIE, Ding N, Meegdes M, Erdkamp F, Heijns JB, Tol J, Vriens BEPJ, Dercksen MW, Aaldering KNA, Pepels MJAE, van de Winkel L, Peters NAJB, van de Wouw AJ, Maaskant SAJG, Teeuwen-Dedroog NJA, van Nijnatten TJA, de Boer M, Tjan-Heijnen VCG. Time trends in real-world treatment patterns and survival in patients diagnosed with de novo HER2+ metastatic breast cancer: an analysis of the SONABRE registry. Breast Cancer Res Treat. 2024 Jun;205(2):287-302. doi: 10.1007/s10549-023-07235-0. Epub 2024 Feb 21. PMID 38381274
- [Result] Lammers SWM, Thurisch H, Vriens IJH, Meegdes M, Engelen SME, Erdkamp FLG, Dercksen MW, Vriens BEPJ, Aaldering KNA, Pepels MJAE, van de Winkel LMH, Peters NAJB, Tol J, Heijns JB, van de Wouw AJ, Teeuwen NJA, Geurts SME, Tjan-Heijnen VCG. The prognostic impact of BMI in patients with HR+/HER2- advanced breast cancer: a study of the SONABRE registry. Breast Cancer Res Treat. 2024 Jan;203(2):339-349. doi: 10.1007/s10549-023-07108-6. Epub 2023 Oct 25. PMID 37878148